CLINICAL TRIAL: NCT07331636
Title: Comparison of Harmoknee Versus Bounding Exercise Protocol on Strength ,Balance ,Agility and Power in Football Players
Brief Title: Comparison of Harmoknee Versus Bounding Exercise Protocol in Football Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0483
Record Dates: First submitted 2025-12-29; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Sports Physical Therapy
Keywords: Harmoknee protocol; Bounding protocol; Football players

STUDY DESIGN:
Intervention Model Description: randomized clinical trial
Who Masked: Outcomes Assessor
Masking Description: assessor will be blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A will be selected randomly and assigned to 8-week Harmoknee exercise program 3 sessions per week, each lasting 45 minutes (5mins warm-up and 5mins cool down) for assessment of strength and balance.
  Interventions: Other: Harmoknee protocol ( Group A )
- Group B (Experimental): Group B will be selected randomly and assigned to 8week Bounding exercise program 3 session per week, each lasting 45 minutes (5mins warm-up and 5mins cool down) for assessment of strength, balance, agility and muscle power.
  Interventions: Other: Bounding protocol ( Group B )

INTERVENTIONS:
Other: Harmoknee protocol ( Group A ) — Group A will be selected randomly and assigned to 8-week Harmoknee exercise program 3 sessions per week, each lasting 45 minutes (5mins warm-up and 5mins cool down) for assessment of strength and balance.
  Arms: Group A
Other: Bounding protocol ( Group B ) — Group B will be selected randomly and assigned to 8week Bounding exercise program 3 session per week, each lasting 45 minutes (5mins warm-up and 5mins cool down) for assessment of strength, balance, agility and muscle power.
  Arms: Group B

SUMMARY:
This is a randomized clinical trial will recruit male football players aged 18-30 years who regularly participated in sports more than 3 years, with a BMI between 18.5-24.9 kg/m².Athletes with smoking habits, those following other specialized training programs, or those taking any drugs that could affect their performance, and had musculoskeletal injury in past 6 months will be excluded. The sample size will be 36 and participants will randomly divided into two groups (18 in each group): Group A: 8-week Harmoknee program, 3 sessions per week (45 minutes each, including warm-up and cool down). Group B: 8-week Bounding program, following the same schedule. The study will measure strength (1RM Test), balance (Star Excursion Test), agility (T-Test), and muscle power (5 Jump Test) at two points: pre-test (before starting) and post-test (after 8 weeks).

DETAILED DESCRIPTION:
Study design: Randomized Clinical Trial Sample size: 36 (18 in each group)

Inclusion Criteria:

* Male football athletes will be included.
* Aged between 18-30 years.
* Minimum 3 years of regular training in sports.
* Athletes containing body mass index between 18.5-24.9kg/m2

Exclusion Criteria:

* Individuals with existing smoking habits.
* Players involved in any training program other than conventional training.
* Athletes having consumption of any drugs that could affect performance.
* History of musculoskeletal injury in past 6 months. Sampling techniques Non-probability purposive sampling technique

Tools:

Muscle strength: 1RM Test(ICC -0.97) Balance: Star excursion Test(ICC -0.95) Agility: T-Test(ICC -0.97) Muscle power: 5 Jump Test(ICC -0.94)

ELIGIBILITY:
Inclusion Criteria:• Male football athletes will be included.

* Aged between 18-30 years.
* Minimum 3 years of regular training in sports.
* Athletes containing body mass index between 18.5-24.9kg/m2

Exclusion Criteria:• Individuals with existing smoking habits.

* Players involved in any training program other than conventional training.
* Athletes having consumption of any drugs that could affect performance.
* History of musculoskeletal injury in past 6 months.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 36 (Actual)
Dates: Start 2025-03-21 (Actual); Primary Completion 2025-10-02 (Actual); Study Completion 2025-11-02 (Actual)

PRIMARY OUTCOMES:
Strength Test: 1 Repetition Maximum | 8 weeks
  The Epley formula is used to estimate a person's 1 Repetition Maximum (1RM)
  1RM=w (1+r/30) After performing warm-up with empty barbell in back squat position for 10 times, athlete can rest for 2 minutes. Then athlete will perform same protocol with addition of 35 pounds weight and goal is to perform maximum repetitions. At final phase, weight (35 pounds) and the maximum repetitions performed by athlete will enter in Epley formula to calculate 1RM of each athlete.
Balance Test: Star Excursion Balance Test | 8 weeks
  The athlete stands on one leg in the center of a star-shaped grid, with lines extending in 8 extending at 45 angle. While balancing on one leg, the athlete uses the other leg to reach along each line as far as possible without losing balance. The maximum reach distance in each direction is recorded. The test is performed on both legs for three times, and the average of multiple trials is taken in centimeters. Calculate the distance in each direction as a percentage by following formula.
  Average distance in each direction (cm) = Reach 1 + Reach 2 + Reach 3 / 3 Relative distance in each direction (%) = Average distance in each direction / leg
Agility Test: T-Test | 8 weeks
  Four cones are arranged in a "T" shape: one at the starting point (Cone A), two at the left and right points (Cones B and C), and one at the top (Cone D).The athlete starts at Cone A and sprints to Cone D (10m).From Cone D, the athlete side-shuffles to Cone B(5m), then across to Cone C(10m), and back to Cone D(5m).Finally, the athlete backpedals from Cone D to Cone A (10m).The time taken to complete the course is recorded. Each athlete completes three attempts, and the best time recorded by stop watch is used for analysis.
Muscle Power Test: 5 Jump Test | 8 weeks
  The athlete starts behind a starting line, standing with both feet shoulder width apart. When ready, they are to perform five consecutive broad jumps non-stop, using a forward as well as a vertical jump style that allows them to gain maximum distance. They are able to use their arms assist the explosive movement and for balance. Paint or any ink will be used under his shoes to mark his steps correctly. The total distance covered after five jumps is measured from the starting line to the point where the athlete lands on the final jump. Each athlete completes two trials, and the best distance is recorded in cm.Rest periods of 1-2 minutes are provided between trials to prevent fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Hadiqa Mishal, DPT, Principal Investigator — Riphah International University
Locations (1):
- Model Town Football Club, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Asimakidis ND, Mukandi IN, Beato M, Bishop C, Turner AN. Assessment of Strength and Power Capacities in Elite Male Soccer: A Systematic Review of Test Protocols Used in Practice and Research. Sports Med. 2024 Oct;54(10):2607-2644. doi: 10.1007/s40279-024-02071-8. Epub 2024 Jul 18. PMID 39026085
- [Background] Wing CE, Turner AN, Bishop CJ. Importance of Strength and Power on Key Performance Indicators in Elite Youth Soccer. J Strength Cond Res. 2020 Jul;34(7):2006-2014. doi: 10.1519/JSC.0000000000002446. PMID 29373431
- [Background] Keiner M, Kadlubowski B, Sander A, Hartmann H, Wirth K. Effects of 10 Months of Speed, Functional, and Traditional Strength Training on Strength, Linear Sprint, Change of Direction, and Jump Performance in Trained Adolescent Soccer Players. J Strength Cond Res. 2022 Aug 1;36(8):2236-2246. doi: 10.1519/JSC.0000000000003807. Epub 2020 Aug 27. PMID 32868678
- [Background] Keller S, Koob A, Corak D, von Schoning V, Born DP. How to Improve Change-of-Direction Speed in Junior Team Sport Athletes-Horizontal, Vertical, Maximal, or Explosive Strength Training? J Strength Cond Res. 2020 Feb;34(2):473-482. doi: 10.1519/JSC.0000000000002814. PMID 30199451
- [Background] Franca C, Gouveia ER, Martins F, Ihle A, Henriques R, Marques A, Sarmento H, Przednowek K, Lopes H. Lower-Body Power, Body Composition, Speed, and Agility Performance among Youth Soccer Players. Sports (Basel). 2024 May 16;12(5):135. doi: 10.3390/sports12050135. PMID 38787004